CLINICAL TRIAL: NCT02816463
Title: Comparison of Oropharyngeal Leak Pressure Between the Ambu AuraGain and the LMA Supreme - a Prospective Randomized Trial
Brief Title: RCT:Oropharyngeal Leak Pressure (OLP) - Ambu AuraGain vs LMA Supreme
Acronym: OLP-Aur/Sup
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, David Wong, Professor, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 14-8360-B
Record Dates: First submitted 2016-06-22; First posted 2016-06-28 (Estimated); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Laryngeal Masks

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ambu AuraGain (Group A) (Experimental): Laryngeal mask Ambu AuraGain will be used, and oropharyngeal leak pressure (OLP) after insertion will be recorded as the primary outcome measure
  Interventions: Device: Ambu AuraGain
- LMA Supreme (Group S) (Active Comparator): Laryngeal mask Supreme will be used, and oropharyngeal leak pressure (OLP) after insertion will be recorded as the primary outcome measure
  Interventions: Device: LMA Supreme

INTERVENTIONS:
Device: Ambu AuraGain
  Arms: Ambu AuraGain (Group A)
Device: LMA Supreme
  Arms: LMA Supreme (Group S)

SUMMARY:
The purpose of this study is to determine whether the leak pressure of the recently introduced laryngeal mask airway, Ambu AuraGain performs superior to the established laryngeal mask LMA Supreme in surgical patients undergoing general anesthesia. This leak pressure is the pressure at which a gas leaks around the airway, which is a key marker of efficacy and safety of its use; a higher leak pressure suggests a better seal between the artificial airway and patient's airway.

ELIGIBILITY:
Inclusion Criteria

ASA physical status I to III Adults more above 18 years Ambulatory surgeries under general anesthesia in supine position requiring laryngeal masks- Knee arthroscopies, bladder tumour resections, hand, eye and general surgical procedures Muscle relaxant not required

Exclusion Criteria

Reduced mouth opening less than 2.5 cms Recent upper respiratory tract infection and sore throat in last 2 weeks Contraindications to laryngeal mask use as in morbid obesity- BMI more than 40 and severe symptomatic esophageal reflux disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2016-06; Primary Completion 2017-05-09 (Actual); Study Completion 2017-05-09 (Actual)

PRIMARY OUTCOMES:
Oropharyngeal leak pressure (OLP) for each airway device after insertion | Within 2-3 minutes after laryngeal mask insertion before start of surgery.
  OLP is defined as 'the anesthesia circuit pressure at which a gas leak occurs around the SAD'.

SECONDARY OUTCOMES:
Phrayngolaryngeal complications | at 1 hr, 2hr and 24 hrs after the surgery
  Complications like sore throat, dysphonia, dysphagia
Postoperative nausea and vomiting (PONV) | at 1 hr, 2hr and 24 hrs after the surgery
  PONV in the post anesthesia care unit (PACU)- PONV will be recorded as only None for No PONV and Yes for present. Severity grading will not be recorded.
Satisfaction of patient and the anesthesiologist with the device | After 1hr in the post anesthesia care unit (PACU)
  Patient satisfaction (5 point scale)- 0 for very dissatisfied to 5 for very satisfied Anesthesiologist satisfaction scale- Low, Moderate and High

CONTACTS AND LOCATIONS:
Overall Officials: David T Wong, MD, Principal Investigator — Uinversity Health Network (UHN), Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wong DT, Ooi A, Singh KP, Dallaire A, Meliana V, Lau J, Chung F, Singh M, Wong J. Comparison of oropharyngeal leak pressure between the Ambu(R) AuraGain and the LMA(R) Supreme supraglottic airways: a randomized-controlled trial. Can J Anaesth. 2018 Jul;65(7):797-805. doi: 10.1007/s12630-018-1120-4. Epub 2018 Mar 26. PMID 29582360